CLINICAL TRIAL: NCT05159869
Title: Meaningful Activity Intervention for Individuals With Early-Stage Dementia: Involving the End User in Intervention Design
Brief Title: User-Led Meaningful Activity and Early-Stage Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00191838; 1K23AG05880901 (Other: National Institute on Aging)
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Dementia
Keywords: Early Stage; well-being; control; neuropsychiatric symptoms; sense of self; cognitive domains; behavioral symptoms
MeSH Terms: conditions — Dementia; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: The third phase of the study will be a pilot randomized controlled trial exploring the design and feasibility of a novel approach to dementia intervention development. Using a two-group randomized, parallel design, 60 persons with dementia will be assigned to treatment (the collaborative creation of a tailored activity plan) or wait-list control. Treatment group participants will receive the intervention, and will be reassessed at 4 months and 12 months from baseline. There will also be a "check-in" after 8 months' time. Four months after their baseline, wait-list controls will receive the same intervention and will be reassessed, and again at 12 months from baseline. There will be an 8-month visit for wait-list controls. This design allows for estimation of effect sizes using a randomized two-group design at four months, confirmation of treatment gains for wait-listed participants from 4-12 months, and evaluation of intervention acceptability.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia. Persons randomized to the User-Led Meaningful Activity intervention group will begin the treatment protocol right after randomization. The intervention will consist of 3-4 sessions lasting 60-90 minutes each in which participants receive feedback from the neuropsychological assessment, identify the basis/topic of the activity plan, receive dementia psychoeducation, and map out an activity gradation plan. There will be a check-in at 8 months. The neuropsychological battery that was administered at baseline will be re-administered 4 months and 12 months after baseline.
  Interventions: Behavioral: User-Led Meaningful Activity Plan
- Wait-List Control (Active Comparator): After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia (i.e., "mild" dementia). Those who meet criteria will be randomly assigned. Persons randomized to the wait-list control group will begin the treatment protocol after four months' time. There will be a check-in at 8 months.The neuropsychological battery that was administered at baseline will be administered 4 months and 12 months after baseline.
  Interventions: Behavioral: User-Led Meaningful Activity Plan

INTERVENTIONS:
Behavioral: User-Led Meaningful Activity Plan — The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression. For example, (1) an individual who is/was a researcher may continue to maintain a job, conduct research, and even publish papers in the early stages of dementia. (2) As the dementia progresses, he or she may be able to continue to run analyses and read/access literature in his or her field. (3) In the moderate stages of dementia, this participant may read his or her existing publications or go to museums showcasing research of interest. As the disease approaches the severe stage, the participant may read very basic books about his or her former profession. (4) In the severe stages of dementia, this study participant may watch videos related to the former profession, e.g., British Broadcasting Corporation (BBC) or National Geographic.

SUMMARY:
Neuropsychiatric symptoms are the most difficult, distressing, and burdensome aspects of dementia care and a catalyst for long-term care placement. Intervention studies have largely focused on helping caregivers manage these symptoms. However, little has been done with regard to persons at the earliest stages of dementia, nor have persons with dementia played a direct and active, central role in helping to design intervention studies. This study focuses on building, pilot testing, and evaluating a tailored activity plan developed with persons with early-stage dementia. The goal of the intervention is to provide persons at this early stage meaningful activities and a plan for adaptation with disease progression.

DETAILED DESCRIPTION:
Dementia, a public health crisis, affects 47.5 million people worldwide and is projected to double in prevalence every 20 years. A degenerative disorder, dementia leads to a decreased ability to communicate and provide for oneself as the disease progresses, which often results in unmet needs. Unmet needs that are associated with dementia include boredom/sensory deprivation, loneliness, and the need for meaningful activity. The inability of persons with dementia to express or fulfill these needs has a range of adverse outcomes, including the manifestation of neuropsychiatric symptoms (NPS, e.g., agitation, aggression). As NPS are the most difficult, distressing, and burdensome aspects of dementia care and a catalyst for long-term care placement, intervention studies have largely focused on helping caregivers manage these symptoms. However, little has been done with regard to persons at the earliest stages of dementia, nor have persons with dementia played a direct and active, central role in helping to design intervention studies.

The lack of involvement of persons with dementia as study partners in the co-construction of interventions results in interventions that may not be relevant to or address the needs of the very population being targeted. Greater involvement of persons with dementia in intervention development is now recognized as a critical strategy for enhancing the relevance, acceptability and reach of interventions. Research suggests that some aspects of the premorbid sense of self are preserved even in advanced stages of dementia. Failure to recognize a person with dementia's continued awareness of sense of self can result in missed opportunities for involvement as a study partner as well as for developing effective therapeutic interventions. Thus, engaging persons with dementia in intervention development in the early stages of the disease can increase the likelihood that interventions are meaningful and linked to a sense of self throughout disease progression.

This study includes persons with early-stage dementia in the development of a meaningful activity plan. Prior activity intervention studies have primarily targeted participants at a moderate or later stage of dementia; consequently, persons with early dementia have largely been underrepresented in this line of research. As meaningful activity is considered central to the well-being of persons with dementia and is known to decrease negative emotions, it is anticipated that activity rooted in the interests and values of persons with early dementia will facilitate well-being as the disease progresses. Consequently, this study evaluates the impact of a co-designed meaningful activity plan via a pilot, two-group randomized trial with a goal of 60 community-dwelling persons with early-stage dementia. Outcomes examined will include well-being, sense of control, frequency and severity of caregiver-reported NPS, sense of self, and cognition.

ELIGIBILITY:
Inclusion Criteria:

Persons with dementia must:

* Be English-speaking
* Have a diagnosis of early-stage dementia based on standard assessments and diagnostic criteria [e.g., Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5)]
* Be medically stable and responsive to the environment (e.g., not comatose). If participants with dementia are on any of four classes of psychotropic medications (antidepressant, benzodiazepines, antipsychotic, or anti-convulsant) or an anti-dementia medication (memantine or a cholinesterase inhibitor), the investigators will require that participants have been on a stable dose for 60 days prior to enrollment (typical time frame in clinical trials) to minimize possible confounding effects of concomitant medications.

Exclusion Criteria:

* Dementia in the moderate or severe stages
* Bed-boundedness, defined as confined to bed or chair for at least 22 hours a day for at least four of the previous seven days
* Are receiving palliative care or are at end-of-life
* A diagnosis of schizophrenia or a bipolar disorder
* Dementia secondary to probable head trauma
* The participant is taking any neuroleptic medications or has any of the following medical diagnosis: (a) restless legs syndrome, (b) delirium, or (c) akathisia, medication-induced, or other movement disorders such as Parkinson's disease or essential tremor.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie G Regier, PhD, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The PI is committed to the open and timely dissemination of research outcomes and will abide by NIH principles for sharing research resources. Plans for resource sharing among the scientific community include presentation and publication of study findings. Constraints imposed by human research subjects protection regulations and the Johns Hopkins University IRB will be recognized as allowed by the NIH. External researchers interested in investigator data, instruments, and other research methodology and procedures will obtain this information through collaborative agreements with the PI, as required by NIH data sharing policy. While the full collected dataset is not available at this time due to its use as preliminary data for follow-up grants, the Data Dictionary, Informed Consent, and Study Protocol are available.

REFERENCES:
- [Background] Regier NG, Hodgson NA, Gitlin LN. Characteristics of Activities for Persons With Dementia at the Mild, Moderate, and Severe Stages. Gerontologist. 2017 Oct 1;57(5):987-997. doi: 10.1093/geront/gnw133. PMID 27986794
- [Background] Cohen-Mansfield J, Thein K, Dakheel-Ali M, Regier NG, Marx MS. The value of social attributes of stimuli for promoting engagement in persons with dementia. J Nerv Ment Dis. 2010 Aug;198(8):586-92. doi: 10.1097/NMD.0b013e3181e9dc76. PMID 20699725
- [Background] Cohen-Mansfield J, Marx MS, Dakheel-Ali M, Regier NG, Thein K, Freedman L. Can agitated behavior of nursing home residents with dementia be prevented with the use of standardized stimuli? J Am Geriatr Soc. 2010 Aug;58(8):1459-64. doi: 10.1111/j.1532-5415.2010.02951.x. Epub 2010 Jun 23. PMID 20579167
- [Background] Regier NG, Gitlin LN. Dementia-related restlessness: relationship to characteristics of persons with dementia and family caregivers. Int J Geriatr Psychiatry. 2018 Jan;33(1):185-192. doi: 10.1002/gps.4705. Epub 2017 Mar 23. PMID 28332736

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 participants with dementia were randomized to the Experimental Group. One of the participants was enrolled to account for possible attrition. 30 Waitlist participants were enrolled. One caregiver (not enrolled) per participant assisted participants in modifying meaningful activities as needed, in accordance with the co-designed plan, based on dementia progression.
Groups:
- Experimental Group - Individuals With Dementia: After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia. Persons randomized to the User-Led Meaningful Activity intervention group will begin the treatment protocol right after randomization. The intervention will consist of 3-4 sessions lasting 60-90 minutes each in which participants receive feedback from the neuropsychological assessment, identify the basis/topic of the activity plan, receive dementia psychoeducation, and map out an activity gradation plan. A brief cognitive screening tool will be administered at six months. The neuropsychological battery that was administered at baseline will be re-administered four months and 12 months later. Follow-up will also involve solicitation of feedback from the person with dementia and his or her caregiver regarding participants' participation in the study.
  User-Led Meaningful Activity Plan: The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression.
- Wait-List Control Group - Individuals With Dementia: After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia (i.e., "mild" dementia). Those who meet criteria will be randomly assigned. Persons randomized to the wait-list control group will begin the treatment protocol after four months' time. The neuropsychological battery administered at baseline will be readministered after four and 12 months.
  User-Led Meaningful Activity Plan: The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression.
Period: Overall Study
Arm/Group | Experimental Group - Individuals With Dementia | Wait-List Control Group - Individuals With Dementia
Started (The number enrolled (61) represents individual participants (individuals with dementia)) | 31 | 30
Caregivers (Not Enrolled) (An additional milestone row has been added to specify the number of individuals with dementia and caregivers within each arm. The Protocol Enrollment number and number of participants started represents the number of individuals with dementia. While an inclusion criterion for study participation was that individuals with dementia had a local caregiver, the intervention targeted individuals with dementia and their outcomes (not caregivers).) | 31 | 30
Individuals With Dementia | 31 | 30
Completed | 31 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected solely for individuals with dementia, the target population for this intervention study. Baseline Characteristics were not collected for caregivers.
Groups:
- Experimental: After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia. Persons randomized to the User-Led Meaningful Activity intervention group will begin the treatment protocol right after randomization. The intervention will consist of 3-4 sessions lasting 60-90 minutes each in which participants receive feedback from the neuropsychological assessment, identify the basis/topic of the activity plan, receive dementia psychoeducation, and map out an activity gradation plan. A brief cognitive screening tool will be re-administered at six months and 12 months. The neuropsychological battery that was administered at baseline will be re-administered 12 months later. Follow-up will also involve solicitation of feedback from the person with dementia and his or her caregiver regarding participants' participation in the study.
  User-Led Meaningful Activity Plan: The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression.
- Wait-List Control: After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia (i.e., "mild" dementia). Those who meet criteria will be randomly assigned. Persons randomized to the wait-list control group will begin the treatment protocol after four months' time. The intervention will consist of 3-4 sessions lasting 60-90 minutes each in which participants receive feedback from the neuropsychological assessment, identify the basis/topic of the activity plan, receive dementia psychoeducation, and map out an activity gradation plan. A brief cognitive screening tool will be re-administered at six months and 12 months. The neuropsychological battery that was administered at baseline will be re-administered 12 months later. Follow-up will also involve solicitation of feedback from the person with dementia and his or her caregiver regarding participants' participation in the study.
  User-Led Meaningful Activity Plan: The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression.
- Total: Total of all reporting groups
Arm/Group | Experimental | Wait-List Control | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.76 (7.028) | 80.30 (6.132) | 79.99 (6.624)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 19 | 20 | 39
  White, Hispanic | 1 | 2 | 3
  Black | 7 | 3 | 10
  Asian | 2 | 3 | 5
  Hispanic/Latino | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Cognitive Function as Assessed by the Wechsler Memory Scale-III
Description: Global cognitive function will be measured by the Wechsler Memory Scale-III (WMS-III) information/orientation subtest, which assesses general personal information and orientation to person, place, and time. Scores range from 0-14, with higher scores indicating more intact global cognitive function. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Wait-List Control: After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia (i.e., "mild" dementia). Those who meet criteria will be randomly assigned. Persons randomized to the wait-list control group will begin the treatment protocol after four months' time.
  User-Led Meaningful Activity Plan: The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression.
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | -0.2 (0.8) | -0.2 (0.9)

2. Primary Outcome: Change in the Cognitive Domain of Attention as Assessed by the Wechsler Adult Intelligence Scale-IV Digit Span Test
Description: Attention will be assessed via the Wechsler Adult Intelligence Scale (WAIS-IV) digit span subtest total score, obtained by adding up the total score on Digit Span Forward, Digit Span Backward, and Digit Span Sequencing. For all 3 tests, range = 0-16, with higher scores indicating better attention. Total raw score range = 0-48. Every series on each digit span subtest consists of two trials, each of which is scored 1 or 0 points. Testing is discontinued when a zero is obtained on both trials of an item. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | 0.6 (0.3) | -0.2 (0.3)

3. Primary Outcome: Change in the Cognitive Domain of Processing Speed as Assessed by the Trail-Making Test Part A
Description: Processing speed will be assessed via the Trail-Making Test Part A. Participants must draw lines connecting 25 numbered circles in sequential order within a maximum time of 150 seconds. The raw completion time in seconds is converted to age-normed T-scores to facilitate standardized interpretation. Lower T-scores indicate slower processing speed, whereas higher T-scores indicate faster processing speed. Regarding clinically relevant thresholds, T-scores are standardized scores with a mean of 50 and a standard deviation (SD) of 10. A T-score below 40 (i.e., 1 SD below the mean) may suggest mild impairment in processing speed. T-scores below 30 (i.e., 2 SDs below the mean) may reflect substantial processing speed dysfunction. T-scores above 60 reflect performance that is above average for the individual's normative peer group. The outcome is measured as a change in T-score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
T-score | 2.6 (6.4) | -0.2 (6.7)

4. Primary Outcome: Change in the Cognitive Domain of Executive Function as Assessed by the Trail-Making Test Part B
Description: Executive function will be assessed via the Trail-Making Test Part B. Participants must draw lines connecting 13 numbered circles alternately with 12 letters of the alphabet, all in ascending order within a maximum time of 300 seconds. The raw completion time in seconds is converted to age-normed T-scores. Lower T-scores indicate potential deficits in executive function, and higher T-scores indicate more intact executive function. For clinically relevant thresholds, T-scores are standardized scores with a mean of 50 and a standard deviation (SD) of 10. A T-score below 40 (i.e., 1 SD below the mean) may suggest mild executive dysfunction. T-scores below 30 (i.e., 2 SDs below the mean) may reflect substantial executive dysfunction. T-scores above 60 reflect above average executive function for the individual's normative peer group. The outcome is measured as a change in T-score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
T-score | 2.7 (7.6) | -0.6 (7.2)

5. Primary Outcome: Change in the Cognitive Domain of Executive Function as Assessed by the Stroop Color-Word Test
Description: Executive function will be assessed via the Stroop Color-Word Test, a 100-item word-color page where word meanings and ink colors are mismatched (score range = 0-100). The participant must name as many correct ink colors as possible within a time limit of 45 seconds. The number of items correctly named is the raw score, which is converted to a T-score based on normative data, with higher T-scores indicating better executive function. For clinically relevant thresholds, T-scores are standardized scores with a mean of 50 and a standard deviation (SD) of 10. A T-score below 40 (i.e., 1 SD below the mean) suggests mild executive dysfunction. T-scores below 30 (i.e., 2 SDs below the mean) suggests substantial executive dysfunction. T-scores above 60 reflect above average executive function for the individual's normative peer group. The outcome is measured as a change in T-score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
T-score | 1.1 (6.9) | 0.4 (5.8)

6. Primary Outcome: Change in the Cognitive Domain of Executive Function as Assessed by the Clock Drawing Test (CLOX1)
Description: Executive function will be assessed via the Clock Drawing Test Part 1 (CLOX 1). Participants will be asked to draw a clock, put in all the numbers, and set the hands to a specific time. The results will be scored using the CLOX method, which specifically evaluates executive function. CLOX1 scores range from 0-15. Lower scores reflect greater impairment. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 1.3 (1.9) | 0.2 (2.2)

7. Primary Outcome: Change in the Cognitive Domain of Immediate Memory and Learning as Assessed by the Repeatable Battery for the Assessment of Neuropsychological Status List Learning Subtest
Description: Immediate memory and new learning will be assessed via the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) subtest of List Learning. In list learning, 10 semantically unrelated words are orally presented to the subject at a two-second rate. The subject is asked to repeat as many words as possible after each of four learning trials. A higher number of words recalled (range 0-40) indicate more intact immediate memory. Raw scores are converted to a scaled score and percentile rank based on normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 2.7 (4.6) | 0.1 (4.4)

8. Primary Outcome: Change in the Cognitive Domains of Memory and Learning as Assessed by the Repeatable Battery for the Assessment of Neuropsychological Status Story Memory Subtest
Description: Memory and new learning will be assessed via the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) subtest Story Memory. Story Memory is a twelve-item short story presented over two trials (score range: 0-24). The story is read aloud at a slow reading speed. After each presentation, the subject is asked to recall as much of the story as he or she can remember, with more items recalled indicating more intact immediate memory. A verbatim criterion is used. Raw scores are converted to a scaled score and percentile rank based on normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 1.8 (3.4) | 0.3 (3.2)

9. Primary Outcome: Change in the Cognitive Domain of Delayed Memory as Assessed by the Repeatable Battery for the Assessment of Neuropsychological Status List Recall Subtest
Description: Delayed memory will be assessed via the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) subtest of List Recall. List Recall requires the participant to remember as many words (range 0-10) from the list learning test as possible after a delay, with a higher number of words recalled indicating more intact delayed recall. Raw scores are converted to a scaled score and percentile rank based on normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 1.2 (2.0) | 0.2 (2.1)

10. Primary Outcome: Change in the Cognitive Domain of Delayed Memory as Assessed by the Repeatable Battery for the Assessment of Neuropsychological Status List Recognition Subtest
Description: Delayed memory will be assessed via the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) subtest of List Recognition. After the List Learning and List Recall tasks (immediate and delayed), the participant is presented with a series of yes/no recognition trials including target words from the original list and foils. One point is awarded for each correct yes/no answer (range = 0-20), with a higher number of words recognized indicating more intact delayed recall. Raw scores are converted to a scaled score and percentile rank based on normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 1.1 (2.3) | 0.2 (2.3)

11. Primary Outcome: Change in the Cognitive Domain of Delayed Memory as Assessed by the Repeatable Battery for the Assessment of Neuropsychological Status Story Memory Subtest
Description: Delayed memory will be assessed via the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) subtest of Story Recall. In Story Recall, participants are asked to recall as many specific details as possible from the story learned in the story memory subtest, with more details indicating more intact delayed recall. Raw scores are converted to a scaled score and percentile rank based on normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 1.4 (3.3) | 0.3 (3.2)

12. Primary Outcome: Change in the Cognitive Domain of Immediate Visual Memory as Assessed by the Rey-Osterrieth Complex Figure Test
Description: Immediate visual (non-verbal) memory will be assessed via the Rey-Osterrieth Complex Figure (ROCF) test. Participants will first copy a complex geometric figure and then immediately reproduce it from memory. Scoring of drawings is based on the widely used 36-point scoring system, with higher scores indicating more intact immediate visual memory. Each of the 18 scoring units is scored based on accuracy and placement criteria. Raw scores are converted to a scaled score and percentile rank based on normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 1.7 (3.8) | 0.4 (3.9)

13. Primary Outcome: Change in the Cognitive Domain of Delayed Visual Memory as Assessed by the Rey-Osterrieth Complex Figure Test
Description: Delayed visual (non-verbal) memory will be assessed via the Rey-Osterrieth Complex Figure (ROCF) test. Participants are asked to draw all the elements of the figure from the initial figure copy that he or she can recall without visual display of the figure. Scoring of drawings is based on the widely used 0-36-point scoring system (score range), with higher scores indicating more intact delayed visual memory. Each of the 18 scoring units is scored based on accuracy and placement criteria. Raw scores are converted to a scaled score and percentile rank based on normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 0.9 (3.4) | 0.2 (3.5)

14. Primary Outcome: Change in the Cognitive Domain of Language as Assessed by the Controlled Oral Word Association Test
Description: Language, specifically verbal fluency, will be assessed via the Controlled Oral Word Association (COWA) test. Participants are asked to come up with as many words as possible that begin with a given letter within a one-minute time period. Participants are also instructed to exclude proper nouns, numbers, and the same word with a different suffix. Score range 0-36. The number of correct responses is totaled, with higher numbers indicating greater verbal fluency, and the sum compared with normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 2.5 (4.3) | 0.4 (4.4)

15. Primary Outcome: Change in the Cognitive Domain of Language as Assessed by the Boston Naming Test
Description: Language will be assessed via the Boston Naming Test (BNT). Participants are asked to name 60 line drawings of objects of graded difficulty, ranging from very common objects to less familiar ones. Objects must be spontaneously named within a 20-second period. If time limit expires, two kinds of prompting cues (one phonemic, one semantic) may be given. Rules allow for discontinuation and for starting the test at an advanced level, thus saving considerable time for subjects without obvious impairment. The examiner will then total the number of spontaneously produced correct responses, the number of cues given, and the number of responses after phonemic cuing and after semantic cuing. Score range 0-60. A higher number of correct spontaneous responses indicates more intact language skills. Scores will be compared to normative data. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Wait-List Control: After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia (i.e., "mild" dementia). Those who meet criteria will be randomly assigned. Persons randomized to the wait-list control group will begin the treatment protocol after four months' time. The neuropsychological battery that was administered at baseline will be re-administered 12 months later.
  User-Led Meaningful Activity Plan: The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression.
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
units on a scale | 2.1 (3.8) | 0.6 (3.9)

16. Primary Outcome: Change in the Cognitive Domain of Language as Assessed by the Repeatable Battery for the Assessment of Neuropsychological Status Semantic Fluency
Description: Language will be assessed via the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) semantic fluency subtest. This test involves the generation of as many unique examples as possible from a given semantic category within 60 seconds. Raw scores typically range from 0 to approximately 30-40, depending on age and clinical status, with higher scores indicating better performance (i.e., greater language fluency and semantic access). The outcome is reported as a change in group mean T2 (4 months) - T1 (baseline), where the raw score is defined as the total number of valid, non-redundant examples generated on the RBANS Semantic Fluency subtest. A positive value indicates improved semantic fluency.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: examples
Groups:
- Experimental: After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia. Persons randomized to the User-Led Meaningful Activity intervention group will begin the treatment protocol right after randomization. The intervention will consist of 3-4 sessions lasting 60-90 minutes each in which participants receive feedback from the neuropsychological assessment, identify the basis/topic of the activity plan, receive dementia psychoeducation, and map out an activity gradation plan. A brief cognitive screening tool will be administered at six months. The neuropsychological battery that was administered at baseline will be re-administered four months and 12 months later. Follow-up will also involve solicitation of feedback from the person with dementia and his or her caregiver regarding participants' participation in the study.
  User-Led Meaningful Activity Plan: The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression.
- Wait-List Control: After participants are recruited, participants will undergo neuropsychological testing prior to randomization in order to establish baseline cognitive functioning and verify that the participants are indeed in the early stages of dementia (i.e., "mild" dementia). Those who meet criteria will be randomly assigned. Persons randomized to the wait-list control group will begin the treatment protocol after four months' time. The neuropsychological battery administered at baseline will be readministered after four and 12 months.
  User-Led Meaningful Activity Plan: The User-Led Meaningful Activity Plan integrates persons with dementia as partners in the co-construction of an intervention involving personally meaningful activity. Activities are graded to correspond with disease progression.
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
examples | 1.5 (3.4) | 0.5 (3.2)

17. Primary Outcome: Change in the Cognitive Domain of Visuospatial Constructional Ability as Assessed by the Rey-Osterrieth Complex Figure Test
Description: Visuospatial constructional ability is assessed using the Rey-Osterrieth Complex Figure (ROCF) test, a neuropsychological task in which participants reproduce a complex geometric figure. Scoring uses the standard 36-point system, in which 18 components are rated for accuracy and placement (0-2 points each). The total raw score ranges from 0 to 36, with higher scores indicating better performance. The outcome is reported as a change in mean raw score from baseline (T1) to 4 months (T2). A positive change score reflects improvement in visuospatial constructional ability.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
points | 1.1 (2.9) | 0.2 (2.9)

18. Primary Outcome: Change in the Frequency x Severity of Neuropsychiatric Symptoms in Persons With Dementia as Assessed by the Neuropsychiatric Inventory (NPI)
Description: Frequency and severity of neuropsychiatric symptoms are measured by the Neuropsychiatric Inventory (NPI) as reported by the primary caregiver. The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as 1 = occasionally, 2 = often, 3 = frequently, 4 = very frequently. Symptom severity is rated as 1= mild, 2 = moderate, 3 = marked. The total score is calculated as a sum of all 12 domain scores and thus ranges from 12 to 144, with a higher score indicating worsening symptoms. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a negative mean indicates an improvement in frequency x severity of symptoms.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | -4.4 (7.32) | -1.0 (7.9)

19. Primary Outcome: Change in the Cognitive Domain of Visuospatial Ability as Assessed by the Repeatable Battery for the Assessment of Neuropsychological Status Line Orientation
Description: Visuospatial ability is assessed using the Line Orientation subtest of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). In this task, participants are asked to match two angled lines to corresponding lines from a semicircular fan of 13 lines. The test includes 10 trials, and each correct match is awarded 2 points, for a total raw score range of 0 to 20. Higher scores indicate better visuospatial performance. The outcome is reported as a change in mean raw score from baseline (T1) to 4 months (T2). A positive score reflects improved visuospatial ability.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
points | 0.4 (2.1) | 0.2 (2.0)

20. Secondary Outcome: Change in Depression as Assessed by the Geriatric Depression Scale
Description: Depression in persons with dementia will be measured by the Geriatric Depression Scale (GDS-15). The GDS-15 is a 15-item self-report scale tested and used extensively with older adults. Scores of 0-4 are considered normal, while scores of 5-8 signify mild depression, 9-11 signify moderate depression, and 12-15 indicate severe depression. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a negative mean indicates an improvement in depressive symptoms.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | -1.3 (2.1) | -0.2 (2.2)

21. Secondary Outcome: Change in Anxiety as Assessed by the Geriatric Anxiety Inventory
Description: Anxiety in persons with dementia will be measured by the Geriatric Anxiety Inventory (GAI). The GAI is comprised of 20 "Agree/Disagree" items designed to assess typical common anxiety symptoms. Scores range from zero (low anxiety) to 63 (high anxiety). The following cutoff scores are supported in the literature: 0-7 (normal anxiety), 8-15 (mild-moderate anxiety), 16-25 (moderate-severe anxiety), and 26-63 (severe anxiety). The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a negative mean indicates an improvement in symptoms of anxiety.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | -2.4 (4.8) | -0.6 (4.7)

22. Secondary Outcome: Change in Sense of Control as Assessed by the MIDI Sense of Control Scale
Description: Sense of control in persons with dementia will be measured by the Sense of Control Scale. This scale has 12 items that measure a person's sense of control over her or his life. Items are scored on a seven-point Likert scale (1=strongly disagree' 2=disagree somewhat' 3=disagree a little' 4=don't know' 5=agree a little, 6=agree somewhat' and 7=strongly agree). Scores range from 12-84, with higher scores indicating greater perceived control. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | 3.6 (6.5) | 0.7 (6.4)

23. Secondary Outcome: Change in Sense of Control as Assessed by the Wallhagen Perceived Control Questionnaire
Description: Sense of control in persons with dementia will be measured by the Wallhagen Perceived Control Questionnaire (PCQ), a 20-item self-report instrument assessing two dimensions of perceived control: (a) Manageability, or belief in one's ability to handle demands, and (b) Goal Attainment, or belief that one can achieve self-set or externally imposed goals. Each item is rated on a 5-point Likert scale from 1 = Strongly Disagree to 5 = Strongly Agree (total score range: 20 to 100, with higher scores indicating greater perceived control). Both the manageability and goal attainment subscales consist of 10 items (score range: 10-50). Subscale scores are summed to compute the total score. The primary outcome is reported as a change score, calculated as T2 (4 months) - T1 (baseline). A positive change score indicates improved perceived control at the group level.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | 3.1 (6.4) | 0.8 (6.3)

24. Secondary Outcome: Change in Sense of Self as Assessed by the Identity-Alzheimer Moderate Test
Description: Sense of self is assessed using the Identity-Alzheimer Moderate (I-AM) Test, where participants complete 20 "I am…" statements. Responses are given orally and recorded by the examiner. Responses are classified using the Watkins et al. (2006) scoring system into four identity categories: idiocentric, small-group, large-group, and allocentric. Stability is measured as the proportion of identity categories present at both T1 (baseline) and T2 (4 months), divided by the total number of unique categories used across both time points (range: 0 to 1). Higher values indicate greater identity stability.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: proportion of identical categories
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
proportion of identical categories | 0.08 (0.18) | 0.01 (0.20)

25. Secondary Outcome: Change in Sense of Self as Assessed by the IMAGE Test
Description: Sense of self in persons with dementia will be measured by the IMAGE test (denoted only by the acronym IMAGE). This test is comprised of 24 descriptive statements, 21 of which refer to the concepts of identity, behavior, and self-satisfaction. Each component contains seven statements belonging to one of seven self-concept domains (moral-ethical, social, personal, physical, family, cognition, emotion). Responses are scored on a four-point Likert scale as follows: 1=totally false, 2=partly false, 3=partly true, and 4=totally true. The total score was obtained by summing all items (minimum score = 24, maximum score = 96), with higher scores indicating more intact sense of self in a given domain. The outcome reported is the mean(SD) of the IMAGE score for each group. The outcome is measured as a change score, calculated as T2 (4 months) - T1 (baseline), whereby a positive mean indicates an improvement in the group mean.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | 3.5 (6.5) | 0.7 (6.4)

26. Other Pre Specified Outcome: Premorbid Cognitive Function as Assessed by the Test of Premorbid Functioning
Description: General intellectual abilities/premorbid cognitive functioning will be assessed via the Test of Premorbid Functioning (TOPF). The TOPF is composed of 70 irregularly spelled words and takes approximately 10 minutes to complete. The participant reads each word aloud. As correct pronunciation of irregular words relies on previously acquired knowledge, it tends to be resistant to brain damage and serves as a proxy for premorbid IQ. The test is discontinued when the participant provides five consecutive incorrect pronunciations. Each correct pronunciation is given a score of 1, and raw scores range from 0-70 with higher scores indicating higher premorbid cognitive function. The raw score is standardized by age and a scaled score is obtained by comparing to the participant's score to normative data based on their demographic classification.
Time Frame: Baseline only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Wait-List Control
Number analyzed (Participants) | 31 | 30
score on a scale | 54.5 (6.2) | 53.1 (5.9)

ADVERSE EVENTS:
Time Frame: From enrollment until follow-up completion, approximately 1 year
Description: Caregivers were not assessed for adverse events
Arm/Group | Experimental | Wait-List Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT05159869/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05159869/SAP_001.pdf